CLINICAL TRIAL: NCT07187154
Title: The Application of Symptoms Management Program Based on the Patient Reported Outcome After Esophagectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NCC3765
Record Dates: First submitted 2023-03-18; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1：Smart Symptom Management Program (Experimental): During the first six months after surgery, patients in the experimental group will use a WeChat mini-program to proactively self-report their symptoms regularly using the Chinese version of the MD Anderson Symptom Inventory for Esophageal Cancer (MDASI-EC). Based on the reported scores and the pre-defined algorithms in the "Post-Esophagectomy Symptom Grading Management Manual", the system will automatically provide personalized self-management guidance for low-grade symptoms. For more severe symptoms, the system will generate alerts to prompt dedicated study nurses to initiate proactive telephone follow-up and provide tailored health coaching.
  Interventions: Device: Smart Symptom Management Program
- Group 2：Routine Care (No Intervention): Patients in the control group will receive standard post-discharge care as per hospital protocol, which includes routine discharge education and instructions to contact the hospital if problems arise. They will not use the WeChat mini-program and will not receive proactive symptom monitoring or coaching calls.

INTERVENTIONS:
Device: Smart Symptom Management Program — During the first six months after surgery, patients in the experimental group will use a WeChat mini-program to proactively self-report their symptoms regularly using the Chinese version of the MD Anderson Symptom Inventory for Esophageal Cancer (MDASI-EC). Based on the reported scores and the pre-defined algorithms in the "Post-Esophagectomy Symptom Grading Management Manual", the system will automatically provide personalized self-management guidance for low-grade symptoms. For more severe symptoms, the system will generate alerts to prompt dedicated study nurses to initiate proactive telephone follow-up and provide tailored health coaching.
  Arms: Group 1：Smart Symptom Management Program

SUMMARY:
1. Research methods Constructed the "Manual for Graded Management of Postoperative Symptoms of Esophageal Cancer" and developed continuous care Procedures.
2. Randomised controlled studies were conducted to verify the effects of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* The patient is aware and able to communicate in Mandarin;
* There are smartphones；
* Proficient in using WeChat mini programs.
* Patients who were scheduled for esophageal cancer resection in participating centers were eligible for inclusion.

Exclusion Criteria:

* Have cognitive impairment or psychiatric illness;
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Postoperative Complications | From the date of surgery until postoperative day 42 (6 weeks).
  The proportion of patients experiencing one or more postoperative complications with a Clavien-Dindo classification of Grade II or higher. Complications will be identified and graded by reviewing patient electronic medical records and discharge summaries. The outcome will be reported as a binary variable (yes/no), and the rate (percentage) will be calculated for each group.
30-Day All-Cause Readmission Rate | From the date of hospital discharge until 30 days post-discharge.
  The proportion of patients readmitted to the hospital for any cause within 30 days of discharge. Data will be confirmed via hospital information system (HIS) records. The outcome will be reported as a percentage.
Mean Score of Symptom Severity Items on the MD Anderson Symptom Inventory (MDASI) Module for Esophageal Cancer | Assessed at baseline (preoperatively), and then at 1 month, 3 months, and 6 months postoperatively
  Symptom severity will be assessed using the symptom severity subscale of the validated MD Anderson Symptom Inventory (MDASI) module for esophageal cancer. This subscale includes 13 core cancer-related symptoms. Patients will rate the severity of each symptom over the last 24 hours on a numeric scale from 0 ("not present") to 10 ("as bad as you can imagine"). The outcome value for each participant at each time point will be the mean score of these 13 symptom severity items. A higher mean score indicates a greater symptom burden.
Mean Score of Symptom Interference Items on the MD Anderson Symptom Inventory (MDASI) Module for Esophageal Cancer | Assessed at baseline (preoperatively), and then at 1 month, 3 months, and 6 months postoperatively
  The impact of symptoms on daily life will be assessed using the symptom interference subscale of the validated MD Anderson Symptom Inventory (MDASI) module for esophageal cancer. This subscale evaluates how symptoms have interfered with 6 different aspects of daily life (e.g., general activity, mood, work) over the last 24 hours. Ratings are on a numeric scale from 0 ("did not interfere") to 10 ("completely interfered"). The outcome value for each participant at each time point will be the mean score of these 6 symptom interference items. A higher mean score indicates a greater negative impact on daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided